CLINICAL TRIAL: NCT01915394
Title: Management of Hospitalized Respiratory Syncytial Virus (RSV) Infected Patients in the Neonatal Intensive Care Unit (NICU) and Control of Epidemics; TurkNICU-RSV Study: A Multicentric, Prospective Trial
Brief Title: Respiratory Syncytial Virus Infection in Neonatal Intensive Care Units Throughout Turkey: Prospective Multicenter Study (TurkNICU-RSV Trial)
Acronym: TurkNICU-RSV
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Serdar Alan, MD, Ankara University
Other Study IDs: TurkNICU-RSV
Record Dates: First submitted 2013-07-26; First posted 2013-08-02 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Syncytial Virus Infections; Infections, Epidemics
Keywords: Respiratory Syncytial Virus Infections; Epidemics; Neonatal Intensive Care Unit; Newborn infants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized Respiratory Syncytial Virus Infected Newborns: All admitted newborns to the neonatal intensive care unit (NICU) will be enrolled in the study

SUMMARY:
The principle purpose of this multicenter trial is to determine the definition, timing and the percentage of nosocomial RSV epidemics throughout Turkey. In addition, secondary purpose of the trial is to determine the prevention strategies of further spread of Respiratory Syncytial Virus (RSV) in the neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed RSV infection with either RSV-strip test or polymerase chain reaction (PCR).
* Admission to the NICU or hospitalized in the NICU between 1 October 2013 and 01 April 2014.

Exclusion Criteria:

* Refused informed consent

Ages: 5 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized RSV infected newborn infants in the NICU.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hospitalized Respiratory Syncytial Virus infected Newborn in the Neonatal Intensive Care Units, and its relation with possible epidemics. | Patients will be followed during hospitalization, with expected average of 3 weeks

SECONDARY OUTCOMES:
Mortality | Patients will be followed during hospitalization, with expected average of 3 weeks
  mortality related to RSV infection and epidemics

CONTACTS AND LOCATIONS:
Overall Officials: Omer Erdeve, MD, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine, Department of Pediatrics, Division of Neonatology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Oncel MY, Mutlu B, Kavurt S, Bas AY, Demirel N, Akyol M, Erdeve O, Dilmen U. Respiratory syncytial virus prophylaxis in preterm infants: a cost-effectiveness study from Turkey. Turk J Pediatr. 2012 Jul-Aug;54(4):344-51. PMID 23692714
- [Background] Dizdar EA, Aydemir C, Erdeve O, Sari FN, Oguz S, Uras N, Dilmen U. Respiratory syncytial virus outbreak defined by rapid screening in a neonatal intensive care unit. J Hosp Infect. 2010 Aug;75(4):292-4. doi: 10.1016/j.jhin.2010.01.013. Epub 2010 Mar 17. PMID 20299133
- [Background] Alan S, Okulu E, Kilic A, Atasay B, Arsan S. Palivizumab use during respiratory syncytial virus outbreak in the neonatal intensive care unit. J Hosp Infect. 2012 Aug;81(4):292-3. doi: 10.1016/j.jhin.2012.05.011. Epub 2012 Jun 20. No abstract available. PMID 22727129